CLINICAL TRIAL: NCT05812508
Title: A Comparative Study Between Bare Scleral Technique and Conjunctival Autograft on Corneal Topography After Pterygium Surgery
Brief Title: Comparison Between Bare Scleral Technique and Conjunctival Auto-graft on Corneal Topography After Pterygium Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Zainab Mahmoud Ali, resident, Sohag University
Other Study IDs: Soh-Med-22-10-02
Record Dates: First submitted 2023-03-04; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Corneal Topography
Keywords: pterygium surgery by bare scleral & autograft
MeSH Terms: interventions — Corneal Topography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pterygium surgery with bare scleral technique: corneal topograghy before and after surgery
  Interventions: Device: corneal topography
- pterygium surgery with conjunctival autograft technique: corneal topograghy before and after surgery
  Interventions: Device: corneal topography

INTERVENTIONS:
Device: corneal topography — corneal topography before and after pterygium surgery by two techniques bare scleral and conjunctival autograft

SUMMARY:
Aim of the work:

To study the corneal topographic pattern changes in patients who have pterygium excision by two surgical techniques (bare sclera, conjunctival autograft).

DETAILED DESCRIPTION:
Pterygium is one of the common ocular surface disorders , it's is an elastotic triangular fibro-vascular tissue covered by conjunctival epithelium that spreads over the cornea. Pterygium causes differences in curvature & power across the cornea .

The prevalence of pterygium varies from 1.1% to 53% globally in different environmental conditions. Risk factors include;UV radiation, geographical latitude near to the equator, outdoor activity , aging, male, and dusty environment.

Pterygium excision is important in patients suffering from blurred vision due to astigmatism . Surgical techniques include ; bare sclera excision, conjunctival autograft, conjunctival transpositional flap, and amniotic membrane grafting. Pterygium excision increases in the mean central corneal curvature & reduces astigmatism that leads to improvement in visual acuity.

Corneal topography is a gold standard in corneal pathology follow-up. Corneal topography is a computer assisted diagnostic tool that creates a three-dimensional map of the surface curvature of the cornea. Corneal topography produces a detailed, visual description of the shape and power of the cornea.

In this study , corneal topography is used to detect how does corneal curvature change after excision of pterygium .

ELIGIBILITY:
Inclusion Criteria:-

* Patients with pterygium not associated with other pathologies (suitable for excision).
* Nasal pterygium extended to the cornea.

Exclusion Criteria: -

* Associated pathologies such as glaucoma, and cataract.
* Corneal opacities or irregularities, scars, dystrophy or ectasia.
* Patients who underwent previous corneal surgery (including refractive surgery)
* Pseudo-pterygium.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pterygium not associated with other pathologies in the eye (suitable for excision) .
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
comparison of topography finding after pterygium surgery by the bare scleral technique. | baseline
  To investigate the corneal topographic changes by imaging the corneal topography before and after pterygium excision (by the bare scleral technique); to detect corneal curvature changes.
comparison of topography finding after pterygium surgery by the conjunctival auto-graft technique. | baseline
  To investigate the corneal topographic changes by imaging the corneal topography before and after pterygium excision (by the conjunctival auto-graft technique); to detect corneal curvature changes.

REFERENCES:
- [Background] Yilmaz S, Yuksel T, Maden A. Corneal topographic changes after four types of pterygium surgery. J Refract Surg. 2008 Feb;24(2):160-5. doi: 10.3928/1081597X-20080201-06. PMID 18297940